CLINICAL TRIAL: NCT06397014
Title: The Clinical Applications of D-type Parastomal Hernia Repair Surgery
Status: Completed | Type: Observational
Sponsor: Daorong Wang (Other)
Responsible Party: Sponsor-Investigator, Daorong Wang, DR, Northern Jiangsu People's Hospital
Organization: Northern Jiangsu People's Hospital (Other)
Other Study IDs: PSH001
Record Dates: First submitted 2024-04-29; First posted 2024-05-02 (Actual); Last update posted 2024-05-02 (Actual); Status verified 2024-04

CONDITIONS: Hernia Repair; Stoma Reconstruction; Function and Appearance

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- D-type
  Interventions: Procedure: D-type stoma lateral hernia repair
- Sugerbaker
  Interventions: Procedure: D-type stoma lateral hernia repair

INTERVENTIONS:
Procedure: D-type stoma lateral hernia repair — underwent D-type stoma lateral hernia repair

SUMMARY:
During the period from February 2018 to February 2022, a study was conducted on patients with parastomal hernia.There were 23 patients who underwent repair surgery for D-type colostomy hernia, while 68 patients underwent traditional laparoscopic repair surgery for hernia.The inclusion criteria were: (1) preoperative diagnosis of parastomal hernia by CT scan; (2) underwent laparoscopic repair surgery or combined laparoscopic repair with abdominal wall and stoma reconstruction surgery.The exclusion criteria were: (1) occurrence of tumor recurrence and/or new tumors during the follow-up period; (2) death or loss to follow-up during the follow-up period.

ELIGIBILITY:
Inclusion Criteria:

(1) preoperative diagnosis of parastomal hernia by CT scan; (2) underwent laparoscopic repair surgery or combined laparoscopic repair with abdominal wall and stoma reconstruction surgery.

Exclusion Criteria:

(1) occurrence of tumor recurrence and/or new tumors during the follow-up period; (2) death or loss to follow-up during the follow-up period.

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: patients with parastomal hernia
Sampling Method: Non-Probability Sample
Enrollment: 91 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2022-02-01 (Actual); Study Completion 2023-08-01 (Actual)

PRIMARY OUTCOMES:
postoperative recurrence rate | 2018-2024
  postoperative recurrence rate
treatment cost | 2018-2024
  treatment cost

CONTACTS AND LOCATIONS:
Locations (1):
- Northern Jiangsu People's Hospital, Yangzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No